CLINICAL TRIAL: NCT01518972
Title: A Placebo-Controlled Trial of Prazosin in Individuals With Co-occurring Alcohol Dependence and PTSD Seeking Abstinence
Brief Title: Prazosin for Alcohol Dependence and Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P20AA017839 (NIH); 1P20AA017839-01 (NIH)
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Abuse; Posttraumatic Stress Disorder
Keywords: Alcohol; Abuse; Use; Disorder; Dependence; Symptoms; Alcoholic; Alcoholism; Prazosin; Drug; Medicine; Medication; Treatment; Study; Placebo; Medical; Management; Craving; Consumption; Binge; Drinking; Drink; Heavy; PTSD; Trauma; Post; Posttraumatic
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Disease; Binge-Eating Disorder; Wounds and Injuries | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prazosin (Experimental): Prazosin medication
  Interventions: Drug: Prazosin
- Placebo (Placebo Comparator): Placebo medication
  Interventions: Drug: Placebo medication

INTERVENTIONS:
Drug: Prazosin — Form: Prazosin will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
  Other Names: Minipress
  Arms: Prazosin
Drug: Placebo medication — Form: Placebo will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the drug prazosin is effective for the treatment of alcohol dependency and symptoms of Posttraumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
Background: Alcohol dependence (AD) is a biologically, genetically based disease, yet the majority of clinically accepted treatments are behaviorally or psychosocially based. PTSD and alcohol use disorders (AUDs) commonly co-occur. This comorbidity is associated with more severe clinical impairment, shorter times to relapse, more treatment recidivism, overall greater use of treatment services, and greater treatment costs.

Neuropharmacology of alcohol and prazosin: Emerging pre-clinical evidence shows that noradrenergic systems are involved in brain processes relevant to AD, such as arousal, reinforcement, and stress responsivity. However, virtually no work to date has attempted to translate this knowledge into clinically effective biological interventions. The investigators have adopted the novel, promising strategy of reducing adrenergic activity by blocking noradrenaline binding to post-synaptic alpha-1 receptors via the non-selective, alpha-1 antagonist, prazosin. Preclinical studies have demonstrated that prazosin decreases reinstatement of alcohol consumption, and preliminary clinical data suggest that prazosin reduces alcohol use in humans with AD and reduces PTSD-related nightmares and other symptoms, though it has not been tested in individuals with comorbid AD and PTSD. Prazosin, FDA approved to treat hypertension, typically has few side effects, and is inexpensive.

Design: Randomized double-blind placebo-controlled clinical trial. Participants: 60 individuals with both AD and PTSD (25% women) with stated goal to abstain from alcohol use.

Intervention: Either prazosin titrated per study protocol or matched placebo for 6 weeks with Medical Management (MM) based on the COMBINE Study procedures and a final study visit two weeks after medication discontinuation.

Measures: The primary outcomes are alcohol use during the 12-week medication phase of the study and reports of craving during the same time period. Daily, prompted Interactive Voice Response (IVR) telephone monitoring will be done throughout the 8-week study to assess the primary outcomes and to provide information on affect and medication adherence. Such daily monitoring provides more accurate reports of alcohol use than standard retrospective outcome measures. Analyses: Hierarchical linear modeling to test for main effects of prazosin+MM versus placebo+MM on alcohol use and PTSD symptoms over time, and to evaluate whether reductions in PTSD mediate the effect of prazosin.

Findings to date: Participants randomized to prazosin had a greater reduction in percent days drinking per week and percent days heavy drinking per week between baseline and week 6 than did placebo participants. No significant differences were detected within or between groups in change from weeks 1 to 6 in total PTSD symptoms. Participants in the prazosin condition reported drowsiness on significantly more days than those in the placebo condition. Public health implications: There is a paucity of safe, tolerable, inexpensive, and efficacious drugs currently available for the treatment of AD and PTSD. Consistent with the extant research evaluating medications for comorbid PTSD/AD, the current evaluation of prazosin also found decreased alcohol consumption but no medication effect on PTSD symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Current primary DSM-IV diagnosis of alcohol dependence(AD)
* Current DSM-IV diagnosis of PTSD
* At least 14 (women) or 21 (men) drinks per week AND at least 2 days of heavy drinking during a consecutive 30 day period in the last 90 days
* Desire to abstain from drinking
* At least 18 years of age
* Good general medical health (see Exclusion Criteria below)
* Capacity to provide informed consent
* English fluency

Exclusion Criteria:

Psychiatric/behavioral:

* psychiatric disorder requiring any medication other than anti-depressants (individuals not on a stable dose of an anti-depressant for at least 30 days prior to randomization will be excluded from the study)
* currently taking disulfiram, acamprosate, or naltrexone in the last 30 days or planning to take any of these medications during the 12-week medication phase of the study
* acutely suicidal or homicidal
* current dependence on any other psychoactive substance other than nicotine or cannabis
* a current diagnosis of opioid abuse, use of any opioid- containing medications, methamphetamines, or benzodiazepines during the previous month, or UDA positive for opioids, methamphetamines, benzodiazepines, or sedative hypnotics

Medical:

* significant acute or chronic medical illness including unstable angina, recent myocardial infarction, history of congestive heart failure, preexisting hypotension (systolic <110) or orthostatic hypotension (defined as a systolic drop > 20mmHg after two minutes standing or any drop with dizziness); insulin-dependent diabetes mellitus; chronic renal or hepatic failure, pancreatitis, Meniere's disease, benign positional vertigo, narcolepsy
* for males only, concomitant use of trazodone (or use in the last 7 days), tadalafil, or vardenafil (or use in the last 3 days) due to increased risk of priapism
* history of prazosin-sensitivity; no prazosin for at least the past 30 days
* women who are pregnant, nursing infant(s), or of childbearing potential and not using a contraceptive method judged by the study physician or PA to be effective
* signs or symptoms of alcohol withdrawal at the time of initial consent
* legal involvement that could interfere with study treatment
* individuals court ordered for treatment will not be eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Simpson, PhD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited from September 2009 to June 2012 (2 years and 9 months). Out of 354 people who inquired about the study, 30 were eligible and randomized.
Pre-assignment Details: Out of 354 individuals who inquired about the study, 54 consented and completed the in-person screen. Out of these 54 individuals, 2 declined participation and 22 were ineligible: 10 individuals did not have PTSD and the rest had an acute illness (4), uncontrolled psychosis (2), legal involvement (2), and other reasons not previously mentioned (4).
Groups:
- Prazosin: Prazosin medication
  Prazosin: Form: Prazosin will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
- Placebo: Placebo medication
  Placebo medication: Form: Placebo will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 15 | 15
Completed | 9 | 11
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Moved from area | 1 | 0
Not completed — Transportation problems | 1 | 0
Not completed — Exclusionary medical condition | 1 | 0
Not completed — Missed safety visits | 0 | 1
Not completed — Exclusionary medication | 0 | 1
Not completed — Declined medication starting on day 12 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study was scaled back from 12 to 6 weeks after enrolling 18 participants because participants had difficulties adhering to a 12-week protocol (54.5 % & 14.3% participants from the Prazosin & Placebo group, respectively, withdrew before week 12). 100% of the Prazosin & 62.5% of the Placebo group completed the study after it was scaled back.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.3) | 43.5 (12.4) | 43.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 4 | 12
  Black | 4 | 8 | 12
  Other | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Number of Drinks per Day, 90 Days Prior to Baseline [Mean (Standard Deviation); unit: drinks per day] — This measurement represents the group's average number of drinks per day, 90 days prior to participants' baseline visit. To get this measurement, in each group, participants' reported daily alcohol consumption was summed and averaged. These averages were then summed and averaged to get the group's average.
  drinks per day | 11 (10.8) | 8.5 (5.1) | 9.75 (8.4)
Total Drinks, 7 Days Prior to Baseline [Mean (Standard Deviation); unit: total drinks per week] — This measurement represents the group's average of total drinks, 7 days prior to participants' baseline visit. To get this measurement, in each group, each participant's self-reported daily alcohol consumption was summed. These aggregates were then summed and averaged to get the group's average.
  total drinks per week | 80.1 (75.1) | 49.6 (44.6) | 64.85 (62.6)
Number of Drinking Days, 7 Days Prior to Baseline [Mean (Standard Deviation); unit: drinking days per week] — This measurement represents the group's average number of drinking days, 7 days prior to participants' baseline visit. To get this measurement, in each group, days of when participants reported some alcohol consumption were summed. These aggregates were then summed and averaged to get the group's average.
  drinking days per week | 5.1 (1.7) | 4.2 (2.8) | 4.65 (2.3)
Baseline Alcohol Craving Score [Mean (Standard Deviation); unit: units on a scale] — This measurement was calculated using the Penn Alcohol Craving Scale (PACS). This questionnaire had 5 questions asking about the frequency, intensity, length, and irresistibility of the participants' craving and their overall average alcohol craving in the week prior to their baseline visit. The rating went from 0 to 6, thus the minimum and maximum possible scores were 0 and 30, respectively. The higher the score, the higher the participants' alcohol craving. Each participant's total score was calculated and then averaged to get the mean craving score of the Placebo & Prazosin groups.
  units on a scale | 22.1 (4.5) | 17.5 (6.8) | 19.8 (6.1)
Baseline PTSD (Post-Traumatic Stress Disorder) Score [Mean (Standard Deviation); unit: units on a scale] — The PTSD score was measured using the PTSD Symptom Scale-Interview Version (PSS-I).
  It had 17 questions asking about how often participants re-experienced, avoided, and aroused by their trauma. The rating went from 0 (not at all) to 3 (5 or more times per week/very much), thus the minimum and maximum possible scores were 0 and 51, respectively. The higher the score, the higher the participants' PTSD score. Each participant's total score was calculated and then averaged to get the mean PTSD score of the Placebo & Prazosin groups.
  units on a scale | 31.5 (8.9) | 31.6 (7.7) | 31.55 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Drinking Days Per Week
Description: Data for this measure came from the Form-42 and daily IVR (Interactive Voice Response) monitoring. The percentage of drinking days of each participant was calculated by summing the number of drinking days and comparing them with the number of total drinking days in the same week. The percentage of drinking days from each week was added and averaged to get the percentage of drinking days per week per participant. The percentage of drinking days of all participants in the Prazosin group was added and averaged to get the mean of the percentage of weekly drinking days of the Prazosin group. These steps were repeated for the Placebo group.
Time Frame: 6 weeks
Population: Percent drinking days per week was examined using multilevel mixed-effects linear regression models with random slope that included treatment group, time, & treatment group x time interaction. Time was modeled as a categorical variable.
Measure: Mean (95% Confidence Interval); unit: percentage of drinking days per week
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 9 | 11
percentage of drinking days per week | 18.1 [-1.1 to 37.4] | 49.3 [31.7 to 66.9]

2. Primary Outcome: Percent Heavy Drinking Days Per Week
Description: Data for this measure came from the Form-42 and daily IVR (Interactive Voice Response) monitoring. Heavy drinking was defined as 5 or more drinks per day for men and 4 or more drinks per day for women. The percentage of heavy drinking days of each participant was calculated by summing the number of heavy drinking days and comparing them with the total number of drinking days in the same week. The percentage of heavy drinking days from each week was added and averaged to get the percentage of heavy drinking days per week per participant. The percentage of heavy drinking days of all participants in the Prazosin group was added and averaged to get the mean of percentage of weekly heavy drinking days of the Prazosin group. These steps were repeated for the Placebo group.
Time Frame: 6 weeks
Population: Percent heavy drinking days per week was examined using multilevel mixed-effects linear regression models with random slope that included treatment group, time, & treatment group x time interaction. Time was modeled as a categorical variable.
Measure: Mean (95% Confidence Interval); unit: Percentage of heavy drinking days/week
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 9 | 11
Percentage of heavy drinking days/week | 3.7 [-14.4 to 21.8] | 27.4 [11.3 to 43.5]

3. Primary Outcome: Total Drinks Per Week
Description: Data for this measure came from the Form-42 and daily IVR (Interactive Voice Response) monitoring. The weekly total drinks of each participant were calculated by adding the number of drinks by week. The total drinks from each week were added and averaged to get the weekly total drinks of each participant. The weekly total drinks of all participants in the Prazosin group were added and averaged to get the total drinks per week for the Prazosin group. These steps were repeated for the Placebo group.
Time Frame: 6 weeks
Population: The total number of drinks per week was examined using multilevel mixed-effects linear regression models with random slope that included treatment group, time, & treatment group x time interaction. Time was modeled as a categorical variable.
Measure: Mean (95% Confidence Interval); unit: drinks per week
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 9 | 11
drinks per week | 7.9 [-15.7 to 31.4] | 27 [5.9 to 48.1]

4. Secondary Outcome: PTSD Symptom Assessments
Description: PTSD symptoms/changes in PTSD (Post-Traumatic Stress Disorder) symptomatology was calculated using data from the IVR (interactive Voice Response) monitoring. PTSD scores were derived by computing the daily average of the item totals for overall PTSD and the symptom clusters. The rating range was 0 (not at all) to 8 (extremely). The higher the score/rating, the more severe the PTSD symptoms. The lowest and highest possible average are 0 and 8, respectively.
Time Frame: 6 weeks
Population: PTSD outcomes between weeks 1 and 6 were analyzed using multilevel mixed-effects linear regression models. Models were adjusted for baseline PTSD severity as measured by corresponding PSS-I scores & sub-scores because measures comparable to the IVR PTSD measures were not available at baseline. Analyses were also adjusted for gender.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 9 | 11
units on a scale
  Total PTSD score | 3.1 [1.9 to 4.2] | 2.5 [1.4 to 3.6]
  Re-experiencing | 3.2 [1.9 to 4.4] | 2.6 [1.4 to 3.8]
  Avoidance/numbing | 2.9 [1.6 to 4.2] | 2.4 [1.2 to 3.6]
  Hypervigilance | 3.2 [2 to 4.4] | 2.4 [1.3 to 3.6]
  Disturbung dreams | 2.5 [1 to 3.9] | 2.8 [1.5 to 4.1]

ADVERSE EVENTS:
Time Frame: The collection of adverse event data started after the first participant was enrolled in early July of 2010. All participants completed their participation by the end of June 2012. Each participant's adverse events were monitored for about 1 to 12 weeks, depending whether they completed the study or not.
Description: Study clinician check participants for adverse events (AE's) on medication day 2, twice weekly during the dose titration phase (days 1-14), & weekly during the continuation phase (days 15-84) through physical examinations, an open-ended question, and an Adverse Symptom Checklist.
  Two participants who were withdrawn by the study staff were excluded, thus there were only 14 total participants/group in the all-cause mortality, serious AE's, and other AE's.
Arm/Group | Placebo | Prazosin
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 14/14 | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Prazosin (N=14)
Experienced 1 adverse event (General disorders) | 2 | 0 — This adverse event can be dizziness on standing, headaches, lightheadedness, nausea, lack of energy, drowsiness, and blood pressure drop from sitting to standing.
Experienced 2 adverse events (General disorders) | 5 | 1 — This adverse event can be dizziness on standing, headaches, lightheadedness, nausea, lack of energy, drowsiness, and blood pressure drop from sitting to standing.
Experienced 3 adverse events (General disorders) | 7 | 9 — This adverse event can be dizziness on standing, headaches, lightheadedness, nausea, lack of energy, drowsiness, and blood pressure drop from sitting to standing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2011-08-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT01518972/ICF_000.pdf